CLINICAL TRIAL: NCT05565560
Title: A Phase 3, Multicenter, Open-label, Single-arm Study to Assess the Efficacy and Safety of Apremilast (AMG 407) in Japanese Pediatric Subjects From 6 Through 17 Years of Age With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Assess the Efficacy and Safety of Apremilast in Japanese Pediatric Participants With Moderate to Severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200346
Record Dates: First submitted 2022-09-20; First posted 2022-10-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Apremilast; AMG 407; Moderate to Severe Plaque Psoriasis; Pediatric Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apremilast (Experimental): Participants with a weight between ≥ 15 kg to < 50 kg will receive apremilast 20 mg twice daily (BID) tablet. Participants weighing ≥ 50 kg will receive apremilast 30 mg BID tablet.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Oral tablets
  Other Names: AMG 407; Otezla

SUMMARY:
The primary objective of this study is to evaluate the efficacy of apremilast in children and adolescents (ages 6 through 17 years) with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants aged 6 to 17 years at screening
* Participants must have a weight of ≥ 15 kg
* Diagnosis of chronic plaque psoriasis for at least 3 months prior to screening
* Has moderate to severe plaque psoriasis at screening and baseline as defined by:
* PASI score ≥ 12; and
* BSA ≥ 10; and
* sPGA ≥ 3 (moderate to severe)
* Disease inadequately controlled by or contraindicated for ≥ 1 topical therapy for psoriasis
* Candidate for systemic therapy or phototherapy

Exclusion Criteria:

* Psoriasis flare or rebound within 4 weeks prior to screening
* Evidence of skin conditions, other than psoriasis, that would interfere with clinical assessments
* Other than psoriasis, history of any clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease
* Prior history of suicide attempt at any time in the participant's lifetime prior to screening or baseline in the study, or major psychiatric illness requiring hospitalization within 3 years prior to signing the assent and informed consent
* Guttate, erythrodermic, or pustular psoriasis at screening and baseline

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
Achievement of a static Physician Global Assessment (sPGA) score of clear (0) or almost clear (1) with at least 2 points reduction from baseline at Week 16 | Week 16

SECONDARY OUTCOMES:
Achievement of at least 75% reduction in Psoriasis Area and Severity Index (PASI) score (PASI-75) from baseline at Week 16 | Baseline, Week 16
Achievement of at least a 50% reduction in PASI score (PASI-50) from baseline at Week 16 | Baseline, Week 16
Percent change from baseline in total PASI score at Week 16 | Baseline, Week 16
Percent change from baseline in affected body surface area (BSA) at Week 16 | Baseline, Week 16
Achievement of Children Dermatology Life Quality Index (CDLQI) (0/1) at Week 16 | Week 16
Change from baseline in CDLQI score at Week 16 | Baseline, Week 16
Number of participants with treatment-emergent adverse events | Approximately 52 weeks
Number of participants with clinically significant changes in vital signs | Approximately 62 weeks
Number of participants with clinically significant changes in laboratory abnormalities | Approximately 62 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (29):
- Japan (29):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu University Hospital, Gifu, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Takagi Dermatological Clinic, Obihiro-shi, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Takeoka Dermatology Clinic, Marugame-shi, Kagawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Saruwatari Dermatology Clinic, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - University of the Ryukyus Hospital, Ginowan-shi, Okinawa
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Nippon Life Hospital, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Sugai Dermatology Park Side Clinic, Utsunomiya, Tochigi
  - St Lukes International Hospital, Chuo-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Mita Dermatology Clinic, Minato-ku, Tokyo
  - Seibo International Catholic Hospital, Shinjuku-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjyuku-ku

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com